CLINICAL TRIAL: NCT05156086
Title: Prospective Study on the Safety and Effectiveness of COVID-19 Vaccine in Kidney Transplant Recipients
Brief Title: Safety and Effectiveness of COVID-19 Vaccine in Kidney Transplant Recipients
Acronym: CoVaKT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jongwon Ha, Professor, Seoul National University Hospital
Other Study IDs: H2110-175-1266
Record Dates: First submitted 2021-12-08; First posted 2021-12-14 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: COVID-19 Vaccination; Renal Transplant
MeSH Terms: interventions — COVID-19 vaccine booster shot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kidney transplant recipients with booster: Patients who received kidney-only transplant or multi-organ transplant including kidney and fully vaccinated with standard dose(s) of messenger RNA (mRNA) or vector vaccine
  Interventions: Drug: COVID-19 vaccine, booster

INTERVENTIONS:
Drug: COVID-19 vaccine, booster — Additional dose of COVID-19 vaccine (booster shot)

SUMMARY:
The current study is a noninterventional prospective study examining the efficacy of additional dosage of the coronavirus disease 2019 (COVID-19) vaccine in kidney transplant recipients (KTRs).

DETAILED DESCRIPTION:
In this clinical, prospective, non-interventional study to assess the effectiveness of an additional dose of COVID-19 vaccination, we evaluated the seroconversion rate of KTRs after the booster shot. Consecutive individuals who have completed standard two-doses of COVID-19 vaccination were enrolled. Following consent, demographic and clinical data were collected from participants, including patient/ transplant characteristics and information regarding previous COVID-19 vaccination.

1 Study visit and sample collection Patients were invited to return for up to 2 follow-up visits for sample collection. Whole blood samples were collected two weeks to 1 day before the booster vaccination and 4 weeks after. During the visit for the second blood sample, a survey was conducted to assess booster-related adverse events.

2. Anti-SARS-CoV-2 antibody assay IgG antibodies against the receptor-binding domain (RBD) of the S1 subunit of the spike protein of severe acute respiratory syndrome coronavirus 2(SARS-CoV-2) were quantified with SARS-CoV-2 IgG II Quant assay (Abbott).

Additionally, neutralizing antibody was assessed using anti-SARS-CoV-2 GenScript cPass SARS-CoV-2 Neutralization Antibody Detection Kit. The cPass detection kit utilizes the horseradish peroxidase (HRP) conjugated recombinant SARS-CoV-2 RBD protein and the human angiotensin-converting enzyme 2 (ACE2) receptor protein. It detects neutralizing antibodies capable of blocking protein interaction between HRP-RBD and ACE2. The assay was performed according to the manufacturer's instructions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who received kidney-only transplantation or multi-organ transplantation including kidney before December 31, 2020
2. Patients ≥ 12 years old
3. Patients fully vaccinated with two standard doses of COVID-19 vaccination with the vector vaccine (AZD1222 of AstraZeneca) or the mRNA vaccines (BNT162b2 of Pfizer-BioNTech or mRNA-1273 of Moderna) including homologous and heterologous regimen.
4. Patients with plans of getting an additional dose of COVID-19 vaccine (i.e., booster shot)
5. Patients providing informed consent and willing to comply with the study protocol, including two blood tests and a survey.

Exclusion Criteria:

1. Patients with a previous history of SARS-CoV-2 infection
2. Who had B-cell depleting therapy (e.g., rituximab, bortezomib) or T-cell depleting therapy (anti-thymocyte globulin) within six months
3. Patients who restarted dialysis due to graft failure

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Kidney transplant recipients fully vaccinated with standard dose(s) of COVID-19 vaccination
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-11-16 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-11-08 (Estimated)

PRIMARY OUTCOMES:
anti-SARS-CoV-2 IgG antibody seroconversion rate | 1 month after booster vaccination
  Seroconversion rate calculated from the anti-SARS-CoV-2 IgG antibody positivity difference before and after the booster shot
adverse event related to booster shot | 1 month after booster vaccination
  local and systemic adverse event related to the third dose of COVID-19 vaccine

SECONDARY OUTCOMES:
Rate of anti-SARS-CoV-2 IgG positivity after standard 2-doses of COVID-19 vaccine | 2week before booster vaccination
Rate of anti-SARS-CoV-2 IgG positivity after additional third doses of COVID-19 vaccine | 1 month after booster vaccination
Change in the quantitative amount of IgG after additional third doses of COVID-19 vaccine | 1 month after booster vaccination
Rate of neutralization antibody positivity after standard 2-doses of COVID-19 vaccine | 2week before booster vaccination
Rate of neutralization antibody after additional third doses of COVID-19 vaccine | 1 month after booster vaccination
Rate of neutralization antibody seroconversion rate upon third doses of COVID-19 vaccine | 1 month after booster vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided